CLINICAL TRIAL: NCT03102580
Title: Patient Osteoarthritis Care Plan To Inform Optimal Treatment
Brief Title: Development of an Osteoarthritis (OA) Care Plan to Improve Process and Quality of OA Treatment Decisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Patricia Franklin, Professor and Director Clinical and Outcomes Research, Department of Orthopedics and Physical Rehabilitation, Northwestern University Feinberg School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHS-1507-31714; PCORI IHS 1507-3174 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2017-01-28; First posted 2017-04-05 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Osteo Arthritis Knee; Osteoarthritis, Hip
Keywords: Shared Decision Making
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Surgeon offices will be randomized to Usual Care or Intervention sites. During Aim 2, after completing the surveys in the clinic, usual care patients and surgeons will have the ability to see PRO scores, but will NOT receive feedback (no OA Care Plan). This is the current standard of care in orthopedic clinics. For intervention sites, the patient and surgeon will receive the OA Care Plan.
  During Aim 3, Usual Care sites will receive the OA Care Plan, and Intervention sites will receive the Enhanced OA Care Plan, including access to Patient Peer Support website and PCP reports (currently under development). All surgeons that used the OA Care plan in Aim 2 will be invited to participate in the Enhanced OA Care plan in Aim 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OA Care Plan Intervention (Experimental): For intervention sites, the patient and surgeon will receive the OA Care Plan (currently under development). The OA Care plan with have Patient Reported Outcomes, feedback reports, and risk factors for shared decision making.
  Interventions: Other: OA Care Plan
- Usual care (No Intervention): As collection of Patient Reported Outcomes (PROs) is considered standard of care in orthopedics (CMS mandate, Bundled Payment requirements, and reporting for Qualified Clinical Data Registry requirement for example), usual care patients and surgeons will have the ability to see PRO scores.

INTERVENTIONS:
Other: OA Care Plan — Patient and surgeon will receive the OA Care Plan (currently under development). This Care Plan will inform Shared Decision for treatment of moderate to sever OA, including surgical and non-surgical options.
  Arms: OA Care Plan Intervention

SUMMARY:
Knee and hip osteoarthritis (OA) is the most common cause of disability in the U.S. and affects more than 60% of adults over 65 years. As the burden of knee and hip OA increases among aging adults, more patients are deciding to have joint replacement surgery. However, no clear guidelines exist for patients to determine if or when to undergo total joint replacement (TJR).

The investigators plan to develop a web-based system that will provide individualized patient OA Care Plans that will help patients make informed decisions about how to treat their arthritis. The investigators will be using this system with patients to see if they find it useful.

The investigators believe that the OA Care plan will improve the process and quality of OA treatment decisions and the quality of OA care.

DETAILED DESCRIPTION:
The investigators propose to prospectively randomize orthopedists, with their patients, to receive (or not) a real-time, web-based system intervention: the OA Care plan. The OA Care plan will include individualized, patient-centric information: (1) trended patient-reported OA pain and function, (2) tailored estimates of likely TJR benefits and risks based on a contemporary US cohort of 25,000 TJR patients (FORCE-TJR Registry), (3) evidence-based information for non-operative care, and (4) individual patient goals.

Specific Aims include:

Aim 1. Patients and their Caregivers/Trusted Others will refine the design, content, and usability of a real-time, web-based individual OA Care plan to guide TJR and non-operative OA care decisions.

Aim 2. Randomize 26 orthopedists, and their patients, to receive the OA Care plan at the time of orthopedic consultation (intervention) vs. usual care (control) and compare (a) OA care decision process and quality and (b) quality of OA care as measured by pain relief and functional gain in the two arms at 6 and 12 months after the decision, and assess the impact of decision quality on quality of OA care.

Aim 3. Randomize 36 orthopedists, and their patients, to receive the OA Care plan plus peer, family, and primary care physician support (OA Care plan+Support; intervention) vs. the OA Care plan alone and compare the quality of OA care decision and quality of care (pain relief, functional gain) in the two arms.

Based on the components of the Chronic Care Model, this technology-delivered, individualized OA Care plan will enable patients and clinicians to make treatment decisions based on patient symptoms, goals, and comparative effectiveness evidence. The investigators hypothesize that OA Care plan users, as compared to usual care, will report greater decision quality for both TJR or non-operative care, and better quality of care (less OA pain, greater function). Further, the investigators anticipate incremental effectiveness of the OA Care plan+Support (peer, family, and primary care support) on the same outcomes. Study results will guide future OA Care plan implementation to assure optimal healthcare for patients with advanced knee and hip OA. Finally, lessons learned from the evaluation of this automated patient-centric decision support system can be extended beyond OA and TJR to other elective surgical procedures to engage informed patients to make optimal individual decisions.

ELIGIBILITY:
Inclusion Criteria:

* All new patients to participating surgeon's practice for the purpose of evaluation of knee or hip OA are possible participants.
* Patients must be 40 years of age or older and able to provide informed consent.

Exclusion Criteria:

* Inflammatory arthritis, such as rheumatoid or psoriatic arthritis
* Recent knee or hip injury as purpose for visit
* Pregnant women
* Prisoners
* Non-English speaking subjects- As we are refining and testing a web-based system intervention that provides individualized patient OA Care plans to improved shared decision making between patients and providers, for research purposes we must assure that the 'counseling' between the surgeon and patient will be in their native language. Once we have identified what materials work at the end of the study, we will translate materials into Spanish.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5713 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia D Franklin, MD MBA MPH, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of doctor-diagnosed arthritis and arthritis-attributable activity limitation--United States, 2010-2012. MMWR Morb Mortal Wkly Rep. 2013 Nov 8;62(44):869-73. PMID 24196662
- [Background] NIH Consensus Statement on total knee replacement. NIH Consens State Sci Statements. 2003 Dec 8-10;20(1):1-34. PMID 17308549
- [Background] Dowsey MM, Nikpour M, Dieppe P, Choong PF. Associations between pre-operative radiographic osteoarthritis severity and pain and function after total hip replacement : Radiographic OA severity predicts function after THR. Clin Rheumatol. 2016 Jan;35(1):183-9. doi: 10.1007/s10067-014-2808-7. Epub 2014 Oct 24. PMID 25339125
- [Background] Nguyen US, Ayers,D.C., Li,W., Harrold L, Franklin PD. Pre-operative Pain and Function: Profiles of Selected TKR Patients among US Surgeons. Amer Coll Rheum 2014.
- [Background] Kurtz SM, Lau E, Ong K, Zhao K, Kelly M, Bozic KJ. Future young patient demand for primary and revision joint replacement: national projections from 2010 to 2030. Clin Orthop Relat Res. 2009 Oct;467(10):2606-12. doi: 10.1007/s11999-009-0834-6. Epub 2009 Apr 10. PMID 19360453
- [Background] Katz JN. Parachutes and Preferences--A Trial of Knee Replacement. N Engl J Med. 2015 Oct 22;373(17):1668-9. doi: 10.1056/NEJMe1510312. No abstract available. PMID 26488698
- [Background] Skou ST, Roos EM, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, Rasmussen S. A Randomized, Controlled Trial of Total Knee Replacement. N Engl J Med. 2015 Oct 22;373(17):1597-606. doi: 10.1056/NEJMoa1505467. PMID 26488691
- [Background] Katz JN. Editorial: appropriateness of total knee arthroplasty. Arthritis Rheumatol. 2014 Aug;66(8):1979-81. doi: 10.1002/art.38688. No abstract available. PMID 24975039
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Cubukcu D, Sarsan A, Alkan H. Relationships between Pain, Function and Radiographic Findings in Osteoarthritis of the Knee: A Cross-Sectional Study. Arthritis. 2012;2012:984060. doi: 10.1155/2012/984060. Epub 2012 Nov 19. PMID 23209900
- [Derived] Stern BZ, Pila S, Joseph LI, Rothrock NE, Franklin PD. Patients' perspectives on the benefits of feedback on patient-reported outcome measures in a web-based personalized decision report for hip and knee osteoarthritis. BMC Musculoskelet Disord. 2022 Aug 23;23(1):806. doi: 10.1186/s12891-022-05764-1. PMID 35999585

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited diverse settings and patients by (1) location, (2) practice type, and (3) patient volume. Thirteen sites and 36 surgeons enrolled 5713 patients. Sites were situated in 11 states, 6 were non-academic sites (50%). Patients were > 40 years of age and provided consent in English or Spanish; had a primary diagnosis of OA in a hip or knee and reported moderate or severe pain or functional limitation on the joint-specific standardized PROs included in the ASK assessment.
Groups:
- OA Care Plan Intervention: For intervention sites, the patient and surgeon received the OA Care Plan with Patient Reported Outcomes, feedback reports, and risk factors for shared decision making.
- Usual Care: As collection of Patient Reported Outcomes (PROs) is considered standard of care in orthopedics (CMS mandate, Bundled Payment requirements, and reporting for Qualified Clinical Data Registry requirement for example), usual care patients and surgeons will view PRO scores as presented in the electronic health record.
Period: Phase 1
Arm/Group | OA Care Plan Intervention | Usual Care
Started | 1764 | 1236
Completed (In this study, Phase 1 and 2 represent 2 separate cohorts. Participants do not flow from Phase 1 to Phase 2.) | 1764 | 1236
Not Completed | 0 | 0
Period: Phase 2
Arm/Group | OA Care Plan Intervention | Usual Care
Started | 2713 | 0
Completed (In this study, Phase 1 and 2 represent 2 separate cohorts. Participants do not flow from Phase 1 to Phase 2.) | 2713 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adults >40 years of age with knee or hip osteoarthritis at initial evaluation by an orthopedic surgeon.
Groups:
- Total: Total of all reporting groups
Arm/Group | OA Care Plan Intervention | Usual Care | Total
Number analyzed (Participants) | 4477 | 1236 | 5713
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (9.2) | 65.7 (9.9) | 66.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2739 | 756 | 3495
  Male | 1738 | 480 | 2218
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 3 | 12
  Asian | 22 | 6 | 28
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 5
  Black or African American | 335 | 93 | 428
  White | 3916 | 1082 | 4998
  More than one race | 88 | 23 | 111
  Unknown or Not Reported | 103 | 28 | 131
Mean OA Pain - Knee/Hip Injury and Osteoarthritis Outcome Score (KOOS/HOOS) [Mean (Standard Deviation); unit: score on a scale] — Baseline pain was assessed using the Knee injury and Osteoarthritis Outcome Score (KOOS) for knee OA patients and the Hip disability and Osteoarthritis Outcome Score (HOOS) for hip OA patients. The HOOS/KOOS is a broadly used 100 point scale (0-100) with 100 reflecting the maximum score and best health status for OA patients. The items are combined into two health domains: Pain and ADL (function/activities of daily living). The pain and ADL domains are scored 0-100 independently (with 100 reflecting the best health status for either pain or ADL). The domains scores are not additive.
  score on a scale | 41.4 (15.5) | 39.3 (16.9) | 41.0 (15.9)

OUTCOME MEASURES:

1. Primary Outcome: Differences in Decision Conflict Scale With ASK vs Usual Care
Description: The Decision Conflict Scale (DCS) is a validated self-report instrument that assesses uncertainty in healthcare decision making. The DCS consists of 16 items, each rated on a 5-point Likert scale. Scores are summed and transformed to a total score from 0 (no conflict) to 100 (high conflict). Lower scores indicate less decisional conflict (better outcome), and higher scores reflect greater decisional conflict (worse outcome). Mean (standard deviation) DCS scores are reported by study arm/group.
Time Frame: 1 month post decision
Population: Patients >40 years of age with knee or hip osteoarthritis and initial evaluation by orthopedic surgeon.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- OA Care Plan Intervention: For intervention sites, the patient and surgeon will receive the OA Care Plan. The OA Care plan with have Patient Reported Outcomes, feedback reports, and risk factors for shared decision making.
  For usual care sites, the patient and surgeon will receive the Patient Reported Outcome Score as is available in the electronic health record.
Arm/Group | OA Care Plan Intervention | Usual Care
Number analyzed (Participants) | 4477 | 1236
Score on a scale | 25.1 (7) | 26.0 (8)

2. Secondary Outcome: Differences in Pain Relief at 6 Months After Enrollment
Description: Pain relief was assessed using the Knee injury and Osteoarthritis Outcome Score (KOOS) for knee OA patients and the Hip disability and Osteoarthritis Outcome Score (HOOS) for hip OA patients. The HOOS/KOOS is a broadly used 100 point scale (0-100) with 100 reflecting the maximum score and best health status for OA patients. The items are combined into two health domains: Pain and ADL (function/activities of daily living). The pain and ADL domains are scored 0-100 independently (with 100 reflecting the best health status for either pain or ADL). The domains scores are not additive.
Time Frame: 6 month followup
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- OA Care Plan Intervention: For intervention sites, the patient and surgeon will receive the OA Care Plan. The OA Care plan with have Patient Reported Outcomes, feedback reports, and risk factors for shared decision making.
  For usual care sites, the patient and surgeon will receive only the routine Patient Reported Outcome score as is available in the electronic health record.
Arm/Group | Usual Care | OA Care Plan Intervention
Number analyzed (Participants) | 1062 | 1554
score on a scale | 20.1 (8.5) | 18.9 (9.1)

3. Secondary Outcome: Difference in Functional Gain at 6 Months
Description: Functional gain was assessed using the Activities of Daily Living (ADL) domain of the Knee injury and Osteoarthritis Outcome Score (KOOS) for knee OA, and the Hip disability and Osteoarthritis Outcome Score (HOOS) for hip OA. The HOOS/KOOS is a broadly used 100 point scale (0-100) with 100 reflecting the maximum score and best health status for OA patients. The items are combined into two health domains: Pain and ADL (function/activities of daily living). The pain and ADL domains are scored 0-100 independently (with 100 reflecting the best health status for either pain or ADL). The domains scores are not additive.
Time Frame: 6 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- OA Care Plan Intervention: For intervention sites, the patient and surgeon will receive the OA Care Plan. The OA Care plan with have Patient Reported Outcomes, feedback reports, and risk factors for shared decision making.
  For usual care sites, the patient and surgeons will receive the Patient Reported Outcome score as is available in the electronic health record.
Arm/Group | OA Care Plan Intervention | Usual Care
Number analyzed (Participants) | 1062 | 1554
score on a scale | 17.1 (8.9) | 18.2 (9.2)

ADVERSE EVENTS:
Time Frame: The 5713 enrolled patients were followed for 12 months.
Groups:
- OA Care Plan Intervention; Usual Care: All enrolled participants were systematically assessed for deaths, serious adverse events, and other adverse events throughout the 12-month study period via patient reports, feedback, and clinical evaluation at regular study visits.
Arm/Group | OA Care Plan Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/4477 | 0/1236
Serious Adverse Events (participants affected / at risk) | 0/4477 | 0/1236
Other Adverse Events (participants affected / at risk) | 0/4477 | 0/1236

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT03102580/Prot_SAP_000.pdf